CLINICAL TRIAL: NCT02484144
Title: Evaluation of the Information of the Patient Before a Scheduled Coronarography
Acronym: INFOCORO
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-04
Record Dates: First submitted 2015-06-24; First posted 2015-06-29 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Cardiac Disease
Keywords: information; coronarography; understanding
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients receive usual information: Patients receive usual information before Scheduled Coronarography
  Interventions: Other: usual information
- patients receive modern information: Patients receive usual information and a information by video before Scheduled Coronarography
  Interventions: Other: modern information; Other: usual information

INTERVENTIONS:
Other: modern information — information by video for coronarography
  Groups: patients receive modern information
Other: usual information — usual information for coronarography

SUMMARY:
French study, multicentrique with the cooperation of several hospital centers . 700 patients (200 in the stage 1 and 500 in the stage 2). Every patient will complete questionnaires in a anonymous way.

DETAILED DESCRIPTION:
Stage 1: evaluation of the score in the population and the evaluation of the improvement of the score after an information more detailed by the educational video.

For that purpose, inclusion on one week with comparison of the score obtained during a classic information with delivery of the sheet of information and during a classic information followed by an information more detailed with educational video.

Check during this stage of the significant improvement of the score with the addition of the educational video literally of information and in the oral information supplied usually within the framework of the current care Evaluation of the number of subject included in the 1 week. Stage 2: Comparison of the patient understanding between 2 groups: 1 group received the information by using the information targeted with educational video (modern information) and the other group the classic information considered as the reference.

Inclusion planned over 2 weeks with for every center 1 week of classic information and 1 week of targeted information, allowing a randomized comparison of the 2 methods.

To limit the biases of inclusions and the effect centers, every center will realize 1 week of every method, according to a specific drawing lots in every center to determine with which information (classic or targeted) the study will begin.

ELIGIBILITY:
Inclusion Criteria:

* hospitalisation for scheduled coronarography

Exclusion Criteria:

* Coronarographies with general anesthesia.
* Patients not speaking or not reading French, or having linguistic knowledge not allowing the delivery of an appropriate information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with scheduled coronarography
Sampling Method: Probability Sample
Enrollment: 821 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Improvement of the quality of the information of the patients | one day
  Improvement of the quality of the information of the patients by a video about the coronarography (realization of the procedure, the profits and the risks) associated with a written information. The quality of the information will be estimated by a dedicated score.

CONTACTS AND LOCATIONS:
Locations (40):
- France (40):
  - CHU Amiens, Amiens
  - CHU Jean MINJOZ, Besançon
  - Chu Avicennes, Bobigny
  - Chu Brest, Brest
  - Hôpital Cardiologique Louis Pradel, Bron
  - Ch Chartres, Chartres
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Chu Mondor, Crétail
  - CHU Dijon, Dijon
  - Chu Grenoble, Grenoble
  - CH Lagny, Jossigny
  - CH MANS, Le Mans
  - Chru Lille, Lille
  - Chu Marseille, Marseille
  - CH, Mâcon
  - CH d'ANNECY-GENEVOIS, Metz-Tessy
  - Groupe intercommunal Le Raincy Montfermeil, Montfermeil
  - CHRU, Montpellier
  - CHI André Grégoire, Montreuil
  - CHU Nord LAENNEC, Nantes
  - Clinique Ambroise Paré, Neuilly-sur-Seine
  - Chu Nimes, Nîmes
  - Chu Pitie Salpetriere, Paris
  - European Georges Pompidou Hospital, Paris
  - Bichat, Paris
  - Chu Ambroise Paré, Paris
  - CHU Saint Antoine, Paris
  - Cochin, Paris
  - Lariboisière, Paris
  - Ch Perpignan, Perpignan
  - Hopital Cardiologique Haut Lévèque, Pessac
  - CHU Poitiers, Poitiers
  - Chu Reims, Reims
  - Chu Rennes, Rennes
  - CH Yves Le FOLL, Saint-Brieuc
  - Centre Cardiologique du Nord, Saint-Denis
  - Chu Strasbourg, Strasbourg
  - CHU Toulouse Rangueil, Toulouse
  - Hôpital Trousseau, Tours
  - CHRU Nancy, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Lattuca B, Barber-Chamoux N, Alos B, Sfaxi A, Mulliez A, Miton N, Levasseur T, Servoz C, Derimay F, Hachet O, Motreff P, Metz D, Lairez O, Mewton N, Belle L, Akodad M, Mathivet T, Ecarnot F, Pollet J, Danchin N, Steg PG, Juilliere Y, Bouleti C; INFOCORO investigators. Impact of video on the understanding and satisfaction of patients receiving informed consent before elective inpatient coronary angiography: A randomized trial. Am Heart J. 2018 Jun;200:67-74. doi: 10.1016/j.ahj.2018.03.006. Epub 2018 Mar 12. PMID 29898851